CLINICAL TRIAL: NCT03383471
Title: A Multicenter, Randomized, Placebo Controlled, Double-blind, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Invossa K Injection in Patients Diagnosed as Knee Osteoarthritis With Kellgren & Lawrence Grade 2
Brief Title: The Efficacy and Safety of Invossa K Injection in Patients Diagnosed With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS-INV-02-3
Record Dates: First submitted 2017-12-11; First posted 2017-12-26 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis
Keywords: chondrocyte cells; osteoarthritis; gene therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invossa K Inj. (Experimental): Invossa K Inj.
  Interventions: Biological: Invossa K Inj.
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Invossa K Inj. — Invossa K Inj.
  Arms: Invossa K Inj.
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intraarticular Invossa K Injection patients diagnosed with Kellgren & Lawrence grade 2 knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 19 and older
2. Patients with IKDC Subjective Knee Evaluation of ≤ 60 of the target knee.
3. Patients with a score of ≥ 40 on the 100 mm pain VAS of the target knee.
4. Patients with grade 2 osteoarthritis as determined by the radiographic criteria of Kellgren and Lawrence
5. BMI should fall between 18.5 and 30
6. Patients who satisfies the clinical/radiational criteria by the American College of Rheumatology guidelines, and applies to one of the following.

   * Age > 50 years old
   * Morning stiffness < 30 minutes
   * Crepitus and Osteophytes
7. With major lesions concentrated in one section of the knee, and with the major lesions considered the main cause of the clinical symptoms
8. Patients with persistent symptoms in spite of conservative therapy for more than 3 months : Improvement of 100 mm VAS are less than 10 mm after 3 months
9. Healthy, with no major findings from the physical examination, hematology, serum chemistry, and urine tests, and no significant medical history
10. Agreed to use an effective contraceptive method during the study period
11. Voluntarily agreed to participate in this study, and signed the informed consent form

Exclusion Criteria:

1. Patients who had been administered with drugs such as oriental medicine, glucosamine and chondroitin within 14 days of baseline visit (But, possible to include after 14 days of wash-out period)
2. Patients taking steroidal anti-inflammatory medications within 14 days of baseline visit (But, possible to include after 14 days of wash-out period)
3. Patients with severe pain in other areas that could effect the diagnosis of the symptoms
4. Patients over Grade 3 osteoarthritis as determined by the radiographic criteria of Kellgren and Lawrence
5. History of surgery like arthroendoscopy within the past 6 months on the target knee
6. Patients who had been administered with immunosuppressants, including antirheumatic drugs (including methotrexate or antimetabolite), within the past 3 months
7. History of injection within the past 3 months on the target knee
8. Pregnant or breastfeeding female
9. With another joint disease apart from degenerative arthritis
10. Patients with hepatitis including carrier
11. Patients with HIV and an infectious disease which is clinically uncontrolled
12. Patients who have any of the following clinically significant diseases or have a medical history within 6 months :

    * Clinically significant heart diseases which are considered by the investigator
    * Uncontrolled hypertension : if the systolic blood pressure exceeds 160 mmHg or diastolic blood pressure exceeds 100 mmHg in a sitting position
    * Kidney disease
    * Liver disease
    * Endocrine disease
    * Uncontrolled diabetes mellitus : HbA1c ≥ 9%
    * Paget's disease, ochronosis, acromegaly, hemochromatosis, Wilson's disease
    * Genetic diseases (hyperkinesia, collagen gene abnormality)
13. Medical history of past or current malignant tumor
14. Patients with a history of anaphylactic reactions
15. Patients with a history of hypersensitivity reactions to the components of this drug, including dimethylsulfoxide, mannitol, dextran 40 or bovine proteins
16. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
17. Patients who administered the INVOSSA K inj.
18. Considered inappropriate by the investigator for participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
IKDC (International knee documentation committee) Subjective Knee Evaluation | Week 0 and 52
  Changes in IKDC Subjective Knee Evaluation (score)
100 mm VAS (Visual analogue scale) | Week 0 and 52
  Changes in 100 mm VAS

SECONDARY OUTCOMES:
WOMAC (The Western Ontario and McMaster Universities Osteoarthritis Index) score | Week 0, 26, 39 and 52
  Changes in WOMAC (score)
IKDC Subjective Knee Evaluation | Week 0, 26 and 39
  Changes in IKDC Subjective Knee Evaluation (score)
100 mm VAS | Week 0, 26 and 39
  Changes in 100 mm VAS
OMERACT-OARSI (Outcome measures in rheumatology-Osteoarthritis research society international) response rate | Week 26, 39 and 52
  OMERACT-OARSI response rate after administration (%)
MRI scan | Week 0, and 52
  Changes in MRI scan
Joint Space Width | Week 0, and 52
  Changes in Joint Space Width (mm)
Biomarker (CTX-I) in blood | Week 0, 26, and 52
  Levels of CTX-I in blood (ng/ml)
Biomarker (CTX-II) in urine | Week 0, 26, and 52
  Levels of CTX-II in urine (ng/ml)
Rescue Medication (Dosage) | Week 0, 4, 12, 26, 39, and 52
  Dosage of Rescue Medication (mg)
Rescue Medication (Frequency) | Week 0, 4, 12, 26, 39, and 52
  Frequency of Rescue Medication (number)
Drop-out rate | Week 0, 4, 12, 26, 39, and 52
  Drop-out rate (%)
Reason of drop-out | Week 0, 4, 12, 26, 39, and 52
  Reason of drop-out is recorded in CRF (Case Report Form), when the patient is dropped-out according to drop-out criteria (e.g. Withdraw a consent, Patients who can not continuously participate in study due to adverse events, Impossible to follow-up of the patient. etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Chul Lee, MD, PhD, Principal Investigator — Department of Orthopedic Surgery, Seoul National University Hospital
Locations (17):
- South Korea (17):
  - Korea University Anam Hospital, Ansan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University School of Medicine, Daegu
  - Chungnam National University School of Medicine, Daejeon
  - Chonnam National University Hwasun Hospital, Hwasun
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - College of Medicine, Hanyang University, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - School of Medicine, Kyung Hee University, Seoul
  - Seoul National University Borame Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea College of Medicine, Seoul
  - Yonsei University School of Medicine, Seoul
  - Ajou University School of Medicine, Suwon